CLINICAL TRIAL: NCT04499300
Title: Elderly Patients and COVID-19 Infection: a Cohort of Fifty Patients Over Ninety Years of Age
Status: Completed | Type: Observational
Sponsor: Murielle Surquin (Other)
Responsible Party: Sponsor-Investigator, Murielle Surquin, Head of geriatry department, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB-COVID-19-90+
Record Dates: First submitted 2020-08-03; First posted 2020-08-05 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Covid positive: Patients over 90 years old hospitalized within the CHU Brugmann between 03/01/2020 and 05/10/2020 with SARS Cov2 infection.
  Interventions: Other: Data collection from medical files
- Sub-group: deceased patients: Patients over 90 years old hospitalized within the CHU Brugmann between 03/01/2020 and 05/10/2020 with SARS Cov2 infection, with death as outcome.
  Interventions: Other: Data collection from medical files
- Sub-group: patients who survived: Patients over 90 years old hospitalized within the CHU Brugmann between 03/01/2020 and 05/10/2020 with SARS Cov2 infection, who survived the infection.
  Interventions: Other: Data collection from medical files

INTERVENTIONS:
Other: Data collection from medical files — Data collection from medical files

SUMMARY:
SARS-CoV2 or CoVid19 disease is a newly described pathology linked to a subtype of the coronavirus family identified in China in December 2019. This pathology can present multiple clinical facets, ranging from asymptomatic forms to more commonly critical pulmonary forms called "Acute Respiratory Distress Syndrome". The elderly population is more at risk for this infection due to the senescence of the immune system, co-morbidities and poly medications. They also often present a greater state of fragility.

This study aims to report the epidemiology of the first 50 patients over 90 years of age hospitalized within the CHU Brugmann hospital.

ELIGIBILITY:
Inclusion Criteria:

* Be over 90 years of age on the date of admission to CHU Brugmann Hospital
* Have a SARS Cov2 infection proven by antigen or RT-PCR on smear and / or typical imaging regardless of the clinical manifestation
* Have been hospitalized at CHU Brugmann between 03/01/2020 and 05/10/2020

Exclusion Criteria:

None

Min Age: 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Same as inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

PRIMARY OUTCOMES:
Demographic data | 5 minutes
  Age, sex, ethnicity
Comorbidities | 5 minutes
  Smoking, Obesity, Diabetes, Arterial hypertension, Coronary pathology, Cerebrovascular disease, chronic renal failure, chronic obstructive pulmonary disease, Neoplasia, Autoimmune disease, Chronic liver disease
Cumulative Illness Rating Scale-Geriatric (CIRS-G) | 5 minutes
  CIRS-G quantifies burden of disease in elderly patients (comorbidity scale). Higher scores indicate higher severity (maximum score = 56 points).
Treatments | 5 minutes
  Under Chronic corticosteroid therapy or Immunosuppressive therapy
Signs and symptoms | 5 minutes
  Presence and date of first apparition: Fever, Cough, Dyspnea, Chest pain, Nausea or vomiting, Diarrhea, Fatigue, Anosmia, ageusia, inappetence, Confusion, Fall, Fracture
Fever | 5 minutes
  Vital signs at hospital admission: Fever
Hypoxemia | 5 minutes
  Vital signs at hospital admission: Hypoxemia
Tachycardia | 5 minutes
  Vital signs at hospital admission:Tachycardia
Hypotension | 5 minutes
  Vital signs at hospital admission: Hypotension
Gasometry | 5 minutes
  Vital signs at hospital admission: Gasometry
Infectious data | 5 minutes
  Contact with confirmed covid person before admission, lives in a retirement home with other cases, Initial bacterial or viral co-infection, Bacterial or viral co-infection during the hospital stay
Blood count | 5 minutes
  Blood count at hospital admission or first recorded
Ionogram | 5 minutes
  Ionogram at hospital admission or first recorded
Liver function | 5 minutes
  Liver function at hospital admission or first recorded
Coagulation | 5 minutes
  Coagulation at hospital admission or first recorded
Renal function | 5 minutes
  Renal function at hospital admission or first recorded
Albumin | 5 minutes
  Albumin at hospital admission or first recorded
CRP | 5 minutes
  CRP at hospital admission or first recorded
Fibrinogen | 5 minutes
  Fibrinogen at hospital admission or first recorded
D-dimers at hospital admission or first recorded | 5 minutes
  D-dimers
NTproBNP | 5 minutes
  NTproBNP at hospital admission or first recorded
CK | 5 minutes
  CK at hospital admission or first recorded
Troponin | 5 minutes
  Troponin at hospital admission or first recorded
Ferritin | 5 minutes
  Ferritin at hospital admission or first recorded
Procalcitonin | 5 minutes
  Procalcitonin at hospital admission or first recorded
Biology - highest rate | 5 minutes
  Highest rate of CRP, D-Dimers, Urea, Creatinin, Fibrinogen, CK, Troponins
Biology - lowest rate | 5 minutes
  Lowest rate of hemoglobin, platelets, leucocytes, lymphocytes, albumin, Na+, K+
Percentage of pulmonary involvement on chest CT scan | 5 minutes
  Percentage of pulmonary involvement on chest CT scan
Number of pulmonary lobes affected | 5 minutes
  Number of pulmonary lobes affected
Type of lesions | 5 minutes
  Type of lesions as reflected on the CT scan images: 'Ground glass' or 'Crazy paving'
Need for oxygenotherapy | 5 minutes
  Need for oxygenotherapy (yes/no)
Means of ventilation | 5 minutes
  Means of ventilation
Treatment received | 5 minutes
  Hydroxychloroquine or Azithromycin
Length of ICU Stay | 5 minutes
  Length of ICU Stay
Status at hospital exit | 5 minutes
  One of the following choices: death, went back home, went back to a retirement home, was placed in a revalidation unit.
Mortality | 5 minutes
  28-day mortality after PCR / CT scan / diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No